CLINICAL TRIAL: NCT05902702
Title: Isotonic Saline for Children With Bronchiolitis - a Randomized Controlled Non-inferiority Trial
Brief Title: Isotonic Saline for Children With Bronchiolitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Slagelse Hospital (Other)
Collaborators: Copenhagen University Hospital at Herlev (Other); Zealand University Hospital (Other); Copenhagen University Hospital, Hvidovre (Other); Holbaek Sygehus (Other); Nordsjaellands Hospital (Other); Nykøbing Falster Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Bronchiolitis project
Record Dates: First submitted 2023-05-31; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Bronchiolitis; Respiratory Disease; Asthma in Children; Viral Infection; Acute Respiratory Infection
Keywords: Nebulized saline; Nasal saline drops; Nasal saline irrigation; Respiratory severity score
MeSH Terms: conditions — Bronchiolitis; Respiration Disorders; Virus Diseases | interventions — Nasal Lavage; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: An investigator-initiated, multicenter, open label, three-arm randomized, controlled non-inferiority trial.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will receive anonymized data for analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nebulized isotonic saline (Experimental): 5 ml of isotonic saline is administered through a nebulizer with a flow of 10 l oxygen/min
  Interventions: Other: Nebulized isotonic saline
- Nasal irrigation with isotonic saline (Experimental): 0.5-2 ml isotonic saline in each nostril administered as nasal drops
  Interventions: Other: Nasal irrigation with isotonic saline
- No treatment with saline (No Intervention): These children will not receive any treatment with isotonic saline, but superficial suctioning of nasal secretions as needed (as part of standard care).

INTERVENTIONS:
Other: Nebulized isotonic saline — The intervention will constitute nebulized isotonic saline.
  Arms: Nebulized isotonic saline
Other: Nasal irrigation with isotonic saline — The intervention will constitute isotonic saline administered as nasal drops.
  Arms: Nasal irrigation with isotonic saline

SUMMARY:
The goal of this randomized clinical trial is to investigate the optimal supportive treatment of bronchiolitis in infants from 0-12 months of age. The main question[s] it aims to answer are:

* To investigate whether isotonic saline should be used as supportive treatment for children with bronchiolitis, and if so, identify the optimal route of administration. The primary outcome is duration of hospitalization.
* To investigate the current epidemiology of the viral pathogens causing bronchitis in children in Denmark, and to assess whether children infected with specific pathogens might benefit from treatment with isotonic saline.

The children are randomized after inclusion through computer randomization to one of the 3 arms in the study:

1. Nebulized isotonic saline
2. Nasal irrigation with isotonic saline
3. No treatment with saline

The investigators will compare treatment with saline (both methods) with no treatment, and the investigators will also compare the two methods of delivery of saline (nebulized vs. nasal irrigation).

DETAILED DESCRIPTION:
Design: An investigator-initiated, multicenter, open label, three-arm randomized, controlled non-inferiority trial.

Study sites: Seven pediatric departments in eastern Denmark (Slagelse Hospital, Holbæk Hospital, Zealand University Hospital Roskilde, Copenhagen University Hospital Hvidovre, Copenhagen University Hospital Herlev, Nordsjaellands Hospital, and Nykoebing Falster Hospital).

Participants: Children aged 0-12 months admitted to a pediatric department or emergency department in eastern Denmark with bronchiolitis, whose parents provide informed consent for participation.

Randomization: Participating children are randomized 1:1:1 through computer randomization to either nebulized isotonic saline, nasal irrigation with isotonic saline or no isotonic saline therapy at all. Participating children will have a nasal sample collected and tested for a panel of viral pathogens. Excess material (1 ml nasal lining fluid) from upper airway respiratory samples will be stored in a research biobank until 31.12.2030 and used for sub-phenotyping of bronchiolitis and for developing personalized treatment and prediction of later asthma by means of host transcriptomics and metabolomics, 16S sequencing of the airway microbiome and meta-transcriptomics.

All other treatment is given according to standard of care guidelines.

Sample size: By including 249 children in total (83 in each arm) the investigators can prove non-inferiority of nasal irrigation or nebulized saline relative to no saline with a non-inferiority limit of 12 hours admission, alpha 2.5% and a power of 80%. The investigators aim to include 300 children in total to account for dropouts.

Recruitment: Children will only be included if both parents provide informed consent.

Perspectives: This study may improve current practice for supportive treatment of children with bronchiolitis. If saline is found to be helpful, it may be implemented into global guidelines. If no effect of saline is found, physicians may stop spending resources and manpower on an ineffective and potentially unpleasant treatment. Second, if saline is effective, but nasal irrigation proves to be non-inferior to nebulization, it may also reduce the workload of nurses, and possibly duration of hospitalization, because the treatment can be delivered by the parents at home. Moreover, the parents are empowered to manage their child's illness themselves, potentially improving the experience of parents as well as the affected child.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0-12 months, whose parents give informed consent to participate, with symptoms of bronchiolitis including at least one of:

  * Runny nose
  * Dry and persistent cough
  * Labored breathing (tachypnea, retractions, nasal flaring)
  * Grunting
  * Cyanosis or apnea
  * Wheezing or crackles on auscultation
  * O2 saturations below 92 %
  * Difficulties feeding

Exclusion Criteria:

* Children with cystic fibrosis or other serious congenital lung diseases
* Children in whom treatment with short-acting beta-2 agonist is initiated (as this is delivered in nebulized isotonic saline).

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Duration of hospitalization | 0-7 days typically (max 14 days)
  In hours

SECONDARY OUTCOMES:
Number of participants needing respiratory support | During admission (up to day 14)
  The need for respiratory support with nasal continuous positive airway pressure or high-flow oxygen therapy.
Number of participants being readmitted after discharge | 30 days after discharge
  If readmitted to the hospital
Respiratory severity score | During admission (up to day 14)
  Respiratory Severity Score with Heart Rate (RSS-HR), scale from 0-12, higher score means worse outcome.
Number of participants needing oxygen therapy | During admission (up to day 14)
  Need for oxygen therapy
Number of participants needing transfer to ICU or SICU | During admission (up to day 14)
  Transfer to the intensive care unit or semi-intensive care unit
Health-related Quality of Life | Up to one month after discharge
  Health-related Quality of Life questionnaire developed by Díez-Gandía et al. (PMID: 34488668) including 12 items. Item responses will be scored using the following algorithm (unweighted method): (1) Each response item will be assigned a value according to its gravity (1 = best level or 9 = worst level). (2) The sum of the scores will be standardized using the min-max normalization to a 0-1-point scale, with 1 indicating the best quality of life and 0 the worst.
Fluid supplements | During admission (up to day 14)
  Requirement of fluid supplements either by nasogastric tube or intravenous
pCO2 | During admission (up to day 14)
  Highest pCO2 measured
Number of participants needing to switch treatment | During admission (up to day 14)
  Clinician-initiated switch to the opposite treatment from the one they were randomized to
Number of participants with visible distress | During admission (up to day 14)
  Visible distress in the child during delivery of treatment
Parents satisfaction | Up to one month after discharge
  Parents satisfaction with the given treatment, questionnaire developed by the investigators exploring satisfaction of 3 items on a scale from 1-10 (total score from 3-30) where higher score means better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Marie M Schoos, MD, PhD, Principal Investigator — Slagelse Hospital

IPD SHARING:
Plan to Share IPD: Yes
We have planned to share all IPD with other researchers upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: We have planned to share all IPD with other researchers upon request 5 years after publication.
Access Criteria: Researchers who request access.

REFERENCES:
- [Derived] Schmidt MN, Daugberg R, Nygaard U, Nielsen XC, Chawes B, Rytter MH, Schoos AM. Normal saline for children with bronchiolitis: study protocol for a randomised controlled non-inferiority trial. BMJ Paediatr Open. 2024 Jan 17;8(1):e002273. doi: 10.1136/bmjpo-2023-002273. PMID 38233083